CLINICAL TRIAL: NCT00107926
Title: Study of Licarbazepine in the Treatment of Manic Episodes of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIC477D2303
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; manic episode; treatment; licarbazepine
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- licarbazepine (Experimental)
  Interventions: Drug: Licarbazepine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Licarbazepine
  Arms: licarbazepine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of an investigational drug for the treatment of manic episodes of bipolar disorder. The investigational drug will be given as additional treatment with either lithium or valproate, which are already FDA (Food and Drug Administration)-approved treatments for mania.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder (type I) with manic or mixed episodes (including patients with/without psychotic features or with/without a history of rapid cycling)
* In need of psychiatric treatment
* Cooperation and willingness to complete all aspects of the study

Exclusion Criteria:

* Current diagnosis other than bipolar I disorder
* History of schizophrenia or schizoaffective disorder
* Drug dependence within 1 month prior to study start or testing positive in a urine drug test
* Suicide attempt within 1 month prior to study start or at immediate risk of harm to self or others
* Any form of psychotherapy within 1 month prior to study start

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2004-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean reduction in manic episodes and major depressive episodes from baseline to endpoint (week 6).

SECONDARY OUTCOMES:
Major improvement in anxiety and depression from baseline to endpoint (week 6)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (12):
  - Investigational Site, La Palma, California
  - Investigational Site, Kansas City, Kansas
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Somerville, Massachusetts
  - Investigational Site, Farmington Hills, Michigan
  - Investigational Site, Staten Island, New York
  - Investigational Site, Madison, Tennessee
  - Investigational Site, Bellaire, Texas
  - Investigational Site, Dallas, Texas
  - Investigational Site, Bellevue, Washington
  - Investigational Site, Kirkland, Washington
  - Investigational Site, West Allis, Wisconsin
- Novartis Investigational Site, Vienna, Austria
- Canada (6):
  - Novartis investigator site, Greater Sudbury
  - Novartis Investigational Site, Kelowna
  - Novartis investigator site, London
  - Novartis investigator site, Montreal
  - Novartis investigator site, Vancouver
  - Novartis investigator site, Verdun
- Colombia (3):
  - Guatemala, Bogotá
  - Guatemala, Medellín
  - Guatemala, Pareira
- Czechia (3):
  - Novartis Investigational Site, Brno
  - Novartis Investigational Site, Hradec Králové
  - Novartis Investigational Site, Prague
- Germany (6):
  - Novartis Investigational Site, Berlin
  - Novartis Investigational Site, Bochum
  - Novartis Investigational Site, Dresden
  - Novartis Investigational Site, Ingolstadt
  - Novartis Investigational Site, Mannheim
  - Novartis Investigational Site, Würzburg
- Novartis Investigational Site, Guatemala City, Guatemala
- Novartis Investigational Site, Lima, Peru
- Russia (2):
  - Novartis Investigational Site, Moscow
  - Novartis Investigational Site, Yaroslavl
- Slovakia (2):
  - Novartis Investigational Site, Bojnice
  - Novartis Investigational Site, Michalovce
- Novartis Investigational Site, Durban, South Africa
- Ukraine (5):
  - Novartis Investigational Site, Dnipro
  - Novartis Investigational Site, Kiev
  - Novartis Investigational Site, Luhansk
  - Novartis Investigational Site, Odesa
  - Novartis Investigational Site, Simferopol
- Novartis Investigational Site, Caracas, Venezuela

REFERENCES:
- See also: Click here for further information and to find an investigational site near you — http://www.novartisclinicaltrials.com/etrials/DiseaseID10/Bipolar-Disorder-clinical-trials.go